CLINICAL TRIAL: NCT03111953
Title: Effect of Biliopancreatic Diversion on Glucose Homeostasis
Acronym: BPD-Mingrone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Catholic University of the Sacred Heart (Other); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 411/14
Record Dates: First submitted 2017-03-13; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Obesity, Morbid
Keywords: Bariatric Surgery; Roux-en-Y gastric bypass; Biliopancreatic Diversion
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGB (Active Comparator): Subjects received Roux-en-Y Gastric Bypass surgery.
  Interventions: Procedure: Roux-en-Y Gastric Bypass Surgery
- BPD (Experimental): Subjects received Biliopancreatic Diversion Surgery
  Interventions: Procedure: Biliopancreatic Diversion Surgery

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass Surgery — In Roux-en-Y Gastric Bypass Surgery a small gastric pouch is created and connected to a segment of jejunum. Bowel continuity is restored by reconnecting the "Roux" limb and the biliopancreatic limb approximately ~75-150 cm distal to the gastrojejunostomy. Therefore, ingested food bypasses most of the stomach, the entire duodenum, and a short segment of the jejunum.
  Arms: RYGB
Procedure: Biliopancreatic Diversion Surgery — In Biliopancreatic Diversion Surgery a horizontal gastrectomy is conducted leaving a portion of the stomach, which is connected to the small intestine, ~250 cm from the ileocecal valve and the biliopancreatic limb is connected to the ileum, ~50 cm from the ileocecal valve. Digestive secretions from the biliopancreatic limb mix in the common channel, where ingested food is also delivered by the alimentary limb.
  Arms: BPD

SUMMARY:
Biliopancreatic diversion (BPD) surgery results in greater resolution of type 2 diabetes than all other bariatric surgical procedures, and it is hypothesized that this procedure has specific beneficial effects on glucose homeostasis beyond weight loss alone. The BPD procedure is performed in more than 150 patients/year by surgeons at the Division of Obesity and Metabolic Disorders, Catholic University of the Sacred Heart, School of Medicine, in Rome, Italy. The purpose of this study is to provide a better understanding of the effect of the BPD bariatric surgical procedure on insulin action and pancreatic beta cell function. It is hypothesized that weight loss achieved with BPD surgery will have greater effects on insulin sensitivity and beta cell function than weight loss induced by Roux-en-Y gastric bypass (RYGB).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 35 kg/m²
* Undergoing either the RYGB or the BPD procedure.
* Able to provide informed consent to participate in the research study

Exclusion Criteria:

* Weight > 450 pounds
* Smoke > 7 cigarettes per day
* Previous malabsorptive or restrictive intestinal surgery
* Pregnant or breastfeeding
* Inflammatory intestinal disease
* Diabetes
* Unstable dose of medications in the last 4 weeks before the pre-surgery metabolic studies
* Severe organ dysfunction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01-09 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in skeletal muscle insulin sensitivity will be assessed using the Hyperinsulinemic-Euglycemic Clamp (HEC) procedure, before and after weight loss induced by either BPD or RYGB surgery | Change from Baseline up to a possible 9 months
  Insulin sensitivity: The HEC procedure will be used to evaluate insulin sensitivity before and after 20% weight loss induced by either BPD or RYGB surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine; Geltrude Mingrone, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angelini G, Salinari S, Castagneto-Gissey L, Bertuzzi A, Casella-Mariolo J, Ahlin S, Boskoski I, Gaggini M, Raffaelli M, Costamagna G, Casella G, Marini PL, Gastaldelli A, Bornstein S, Mingrone G. Small intestinal metabolism is central to whole-body insulin resistance. Gut. 2021 Jun;70(6):1098-1109. doi: 10.1136/gutjnl-2020-322073. Epub 2020 Sep 29. PMID 32994312
- [Derived] Harris LA, Kayser BD, Cefalo C, Marini L, Watrous JD, Ding J, Jain M, McDonald JG, Thompson BM, Fabbrini E, Eagon JC, Patterson BW, Mittendorfer B, Mingrone G, Klein S. Biliopancreatic Diversion Induces Greater Metabolic Improvement Than Roux-en-Y Gastric Bypass. Cell Metab. 2019 Nov 5;30(5):855-864.e3. doi: 10.1016/j.cmet.2019.09.002. Epub 2019 Oct 3. PMID 31588013